CLINICAL TRIAL: NCT07156708
Title: Effects of Aquatic Aerobic Exercises Combined With Cognitive Tasks on Cognitive Function and Other Health-related Outcomes in Older Adults
Brief Title: Aquatic Exercises Combined With Cognitive Tasks for Older Adults
Acronym: WaterCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90526525.0.0000.5313
Record Dates: First submitted 2025-08-26; First posted 2025-09-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: Physical exercise; Physical activity; Dual-task training; Water-based exercise; Cognitive function; Physical fitness; Mental health; Sleep quality; Quality of life; Cardiovascular parameters
MeSH Terms: conditions — Motor Activity; Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This trial is a randomized clinical trial employing a 1:1:1 allocation ratio. It was designed as a superiority trial with three parallel groups and blinded to outcome assessors and data analysis.
Who Masked: Outcomes Assessor
Masking Description: Blinding is applied to outcome assessors and data analysts responsible for evaluating both primary and secondary outcomes. However, due to the nature of the interventions, blinding is not feasible for the staff conducting the exercise sessions or the participants. To maintain assessor blinding, participants are instructed not to disclose their group allocation or discuss intervention details during outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquatic aerobic exercise program combined with cognitive tasks (Experimental)
  Interventions: Other: Aquatic aerobic exercise program; Other: Cognitive tasks
- Conventional aquatic aerobic exercise program (Experimental)
  Interventions: Other: Aquatic aerobic exercise program
- Control group (No Intervention)

INTERVENTIONS:
Other: Aquatic aerobic exercise program — The aquatic exercise sessions include the following exercises: butt kick, frontal kick, cross-country skiing, and stationary running. These exercises are commonly used in water aerobics classes and provide controlled osteoarticular impact, being safe for older women (Alberton et al., 2019). Training intensity is prescribed using Borg's 6-20 rating of perceived exertion (RPE) scale. The adopted strategy is based on interval training, which alternates between high-intensity effort and low-intensity active recovery phases. Each block consists of 4 minutes of effort (RPE 13 - 15), with one minute for each exercise (butt kick, frontal kick, cross-country skiing, and stationary running) followed by 1 minute of active recovery (RPE 11), performed with stationary running. To facilitate monitoring, an RPE scale (measuring 0.90 × 1.20 m) is fixed to the outside of the pool, in front of the participants.
  Arms: Aquatic aerobic exercise program combined with cognitive tasks; Conventional aquatic aerobic exercise program
Other: Cognitive tasks — This group performs the same aerobic training protocol used by the conventional aquatic program group. Additionally, cognitive tasks are performed during the active recovery phases. Cognitive training encompasses different domains of cognition in all sessions, including semantic fluency, processing speed, cognitive flexibility, inhibitory control, memory, attention, and reasoning. The exercises vary in each class, with progression in complexity in each mesocycle.
  Arms: Aquatic aerobic exercise program combined with cognitive tasks

SUMMARY:
The aquatic environment has characteristics that favor the adherence of older adults to exercise programs, and studies have shown that programs in this setting are effective in enhancing various aspects of physical fitness as well as cognitive function in this population. Research has explored whether incorporating cognitive tasks into an aquatic exercise program could offer additional benefits, but it remains uncertain whether this approach leads to greater improvements in cognitive function compared to aquatic exercises alone. The present protocol reports the WaterCog Study, which aims to evaluate the effects of an aquatic aerobic exercise program combined with cognitive tasks, compared to a conventional aquatic aerobic exercise program and a control group, on cognitive function and other health-related outcomes in older adults. This trial is a randomized, single-blinded, three-arm, parallel, superiority trial. A total of 98 older adults are randomized into one of three groups: 1) an aquatic aerobic exercise program combined with cognitive tasks, 2) a conventional aquatic aerobic exercise program, and 3) a control group. Participants in both exercise groups complete a 12-week exercise program with two weekly sessions on non-consecutive days. The primary outcome is cognitive function, while secondary outcomes include physical function, cardiovascular, and psychosocial parameters. Outcomes are measured at baseline, post-intervention, and at the 12-week follow-up after the end of the intervention period. The analysis plan will employ an intention-to-treat approach and per-protocol criteria. The conceptual hypothesis of the study is that both training programs will significantly improve the investigated outcomes compared to the control group. Additionally, it is expected that aquatic exercises with cognitive tasks will promote additional benefits in cognitive function, with similar gains in physical function, cardiovascular, and psychosocial parameters compared to conventional aquatic aerobic exercises in post-intervention and follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* Older women aged 60 and 75 years;
* Being physically inactive, meaning not participating in physical exercise for at least six months (regular exercise is defined as engaging in any physical training for a minimum of 20 minutes on two or more days a week).

Exclusion Criteria:

* History of cardiovascular disease (except controlled hypertension);
* Osteoarticular limitations for the practice of exercises;
* Being illiterate due to the self-completion questionnaires and the characteristics of the intervention;
* Diagnosis of dementia, schizophrenia, or major depressive disorder.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Objective cognitive function - Digit Span Test | Baseline (week 0), post-intervention (week 13), and 12-week follow-up (week 25)
  The Digit Span Test is used to assess working memory and attention span (Schroeder et al., 2012). The Digit Span Test requires participants to verbally recall a sequence of numbers dictated by the examiner. The test begins with three numbers ranging from 0 to 9, read at 1-second intervals, which participants must remember in the correct order. The sequence increases by one digit if pronounced correctly. If participants fail to recall the correct sequence twice in a row, the test ends. The number of digits correctly recalled is recorded as the test result, with a higher score indicating better performance.
Objective cognitive function - Controlled Oral Word Association Test | Baseline (week 0), post-intervention (week 13), and 12-week follow-up (week 25)
  The Controlled Oral Word Association Test (COWAT) is used to assess verbal fluency, working memory, and inhibitory control (Ross et al., 2007). In this test, participants must say as many words as possible that start with the letters "F," "A," and "S" within 1 minute for each letter. Proper names, repeated words, and variations in gender, number, and conjugation are not considered. A higher number of words in each test indicates better verbal fluency.

SECONDARY OUTCOMES:
Objective cognitive function - Trail Making Test (TMT) | Baseline (week 0), post-intervention (week 13), and 12-week follow-up (week 25)
  The validated version of the Trail Making Test (TMT) for the Brazilian population is used to assess aspects of objective cognitive function (Carvalho & Caramelli, 2020). In the first part of the instrument (TMT-A), which measures visual attention and processing speed, participants must draw a line connecting the numbers 1 to 25 in ascending order. In the second part (TMT-B), which measures cognitive flexibility and executive function, participants connect numbers (1-13) and letters (A-L) in an interleaved numerical and alphabetical order. Participants are instructed to maintain pencil-and-paper contact throughout the test, and shorter completion times indicate better performance.
Self-perception of cognitive function | Baseline (week 0), post-intervention (week 13), and 12-week follow-up (week 25)
  The Brazilian version of the Cognitive Failures Questionnaire (CFQ) is used to measure the frequency of cognitive failures in everyday life, such as lapses in attention, memory problems, and failures in executing intentional actions (Paula et al., 2017). The questionnaire consists of 25 self-administered items, with responses on a Likert-type scale from 0 to 4, which assess the frequency of cognitive failures in different everyday contexts. The total score ranges from 0 to 100 points, with higher scores indicating a greater perceived frequency of cognitive failures and, therefore, poorer self-perception of cognitive function.
Aerobic fitness | Baseline (week 0) to post-training (week 13)
  The 6-minute Walk Test (6MWT) is performed to measure aerobic fitness. The course proposed in the original test is 45.72 m rectangular. The course will be adapted for a straight line of 30 m in length, demarcated with cones every 3 m. Participants are instructed to walk for 6 minutes in a flat 30m course, where the total distance walked "as fast as possible" is assessed
Lower limb strength | Baseline (week 0) to post-training (week 13)
  The 30-s Chair-Stand test is performed to measure the strength of the lower limbs. Participants are instructed to sit and stand up from a chair 43 cm high from the seat, without the aid of the upper limbs, as many times as possible for 30 s. The total number of complete repetitions performed within the 30 seconds is recorded as the result, with higher values indicating greater lower body strength.
Upper limb strength | Baseline (week 0) to post-training (week 13)
  The Arm Curl test is performed to measure the strength of the upper limbs. Starting at full elbow extension and holding a 2 kg dumbbell in each hand, participants are instructed to perform the maximal number of elbow crunches over the full range of motion for 30 s. The test is performed with both upper limbs. The total number of complete repetitions performed within the 30 s is recorded as the result, with higher values indicating greater upper body strength.
Lower limb flexibility | Baseline (week 0) to post-training (week 13)
  The Sit-and-Reach test is performed using a Wells Bench to assess lower limb flexibility, particularly of the hamstring and lower back muscles. Participants sit barefoot on the floor with their legs extended and together, knees fully extended, and the soles of the feet flat against the front of the bench. With arms extended and hands overlapping, they slowly bend forward from the hips, sliding their hands along the measurement scale on the bench, without flexing the knees or using compensatory movements. The maximum reach is held for approximately two seconds, and the greatest distance reached in centimeters in three attempts is recorded.
Agility and dynamic balance | Baseline (week 0) to post-training (week 13)
  The Timed Up and Go (TUG) test is performed to measure agility and dynamic balance. Participants are instructed to get up from the chair (43 cm), turn around a marker that will be 3m, and return to the starting position. The shortest time of the two attempts is considered the result.
Dual-task performance | Baseline (week 0) to post-training (week 13)
  Dual-task performance involves simultaneously performing the TUG test and a cognitive task. Participants are instructed to do the TUG while reciting alternating letters (e.g., A, C, E, etc.). The time taken for the TUG and the number of correctly recited letters are recorded as test results.
Blood pressure | Baseline (week 0) to post-training (week 13)
  Office systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurements are obtained using calibrated and automated oscillometric devices (HEM-7320, OMRON, China). Participants are kept in a calm environment for 5 min, and then measurements are performed in both arms of the participant. Three measurements, with an interval of 1 to 2 min, are taken in the arm with the highest initial value. The average of the three measurements is considered the subject's office blood pressure.
Blood pressure reactivity | Baseline (week 0) to post-training (week 13)
  Blood pressure reactivity is measured as the difference between values recorded during a mental stressor and those obtained at rest. The Stroop Test (Stroop, 1935) is used to induce mental stress, presented via a video on a screen in front of the participant for three minutes. Every two seconds, a visual stimulus consisting of a word written in a specific color will appear, with the color of the word and its meaning being incongruent (for example, the word "blue" written in red). The participant must respond verbally and as quickly as possible to the color of the letters, ignoring the meaning of the word.
  Throughout the test, systolic and diastolic blood pressure are measured by the auscultatory method, using a stethoscope and a calibrated aneroid sphygmomanometer, with one reading every minute, for a total of three readings. The reference arm is the same one used for resting BP assessments. After completing the test, participants are asked to rate their perceived stress level using a
Heart rate variability | Baseline (week 0) to post-training (week 13)
  Heart rate variability (HRV) is measured with participants seated and resting for 10 minutes, during which time their heart rate is continuously recorded using the Polar H10 chest sensor, a validated and widely used device for HRV analysis. Data collection takes place in a quiet environment, with a controlled temperature between 24°C and 26°C. Data is collected via Bluetooth and stored in the Polar Flow app, later exported in a compatible format (.txt or .csv). The final five minutes of the resting period are considered for analysis, as they offer greater physiological stability. Data are processed in Kubios HRV® software, with automatic artifact correction using a low threshold filter. HRV analysis follows the recommendations of the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology (1996), considering time-domain parameters such as SDNN (Standard Deviation of NN Intervals), which reflects the global variability of autonomi
Depressive and anxiety symptoms | Baseline (week 0) to post-training (week 13)
  The validated version of the HADS for the Brazilian population is used to assess depressive and anxious symptoms (Botega et al., 1995). It is an instrument composed of 14 items, seven of which form the anxiety subscale and the other seven the depression subscale, allowing the assessment of symptoms in the previous week. Each HADS item has four response options ranging from 0 to 3, reaching a maximum of 21 points in each subscale. Participants are instructed to answer the questions based on the last 7 days. Based on the final score of each subscale, participants are categorized as having symptoms of anxiety or depression as "unlikely" (0 to 7 points), "possible" (8 to 11 points), and "probable" (12 to 21 points). Higher scores indicate more severe symptoms and a worse perceived emotional state.
Sleep quality | Baseline (week 0) to post-training (week 13)
  The validated version of the Pittsburgh Sleep Quality Index (PSQI) for the Brazilian population is used to assess subjective sleep quality and related disorders (Bertolazi et al., 2011). The questionnaire consists of 19 items, grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping medications, and daytime dysfunction. Each component is scored from 0 (no difficulty) to 3 (severe difficulty), and the sum of the scores results in an overall score ranging from 0 to 21; scores greater than 5 indicate poor sleep quality.
Self-reported quality of life | Baseline (week 0) to post-training (week 13)
  Quality of life is assessed using the WHOQOL-BREF questionnaire, developed by the World Health Organization and previously validated in the Brazilian population (Fleck et al., 2000). The WHOQOL-BREF comprises 26 items divided into four domains: physical, psychological, social relationships, and environment. This instrument is self-administered, with a 5-point Likert scale, and produces standardized scores ranging from 0 to 100, with higher values indicating better perceived quality of life.

OTHER OUTCOMES:
Cognitive status | Baseline (week 0)
  The validated version of the Mini-Mental State Examination (MMSE) (Brucki et al., 2003) for the Brazilian population is used to screen for cognitive decline, and in this study, it is also used to stratify randomization. The questionnaire is divided into two sections: the first, with a maximum score of 21, requires vocal responses regarding temporal and spatial orientation, memory, and attention; the second, with a maximum score of 9, assesses the ability to name, follow commands, write, and copy a polygon. The maximum total score is 30 points, and the test is not timed. Participants' cognitive function is classified based on cutoff points adjusted for education, as proposed by Brucki et al. (2003). The score is formed by the sum of the items answered correctly; the higher the score, the better the cognitive function.
Sociodemographic and clinical characteristics | Baseline (week 0)
  Sociodemographic data, health history, medical conditions, and medication use are collected using a standardized questionnaire before the intervention.
Body mass | Baseline (week 0) to post-training (week 13)
  Body mass measurements are performed using a digital scale with a stadiometer (Welmy, Santa Bárbara d'Oeste - São Paulo, Brazil). Body mass is measured in kilograms.
Height | Baseline (week 0) to post-training (week 13)
  Height measurements are performed using a digital scale with a stadiometer (WELMY, Santa Bárbara d'Oeste - São Paulo, Brazil). Height is measured in meters.
Body mass index (BMI) | Baseline (week 0) to post-training (week 13)
  The calculation of the BMI is performed using the equation: BMI = body mass (kg)/height² (m).
Waist and hip circumferences | Baseline (week 0) to post-training (week 13)
  Waist and hip circumferences are measured with a measuring tape placed around the navel height and the width of the participants' hips, respectively, to calculate the waist-hip ratio.
Physical activity levels | Baseline (week 0) to post-training (week 13)
  The self-reported physical activity level is measured at baseline and post-intervention using the Godin-Shephard Leisure-Time Physical Activity Questionnaire. The translated and validated Brazilian version of the Godin-Shepard questionnaire is used (São-João et al., 2013). Participants should report the number of times they perform vigorous, moderate, and light physical activities for more than 15 minutes a week. The weekly frequencies of intense, moderate, and light activities should be multiplied by nine, five, and three, respectively. The total weekly leisure activity is calculated in arbitrary units from the sum of the products of each component, allowing for categorizing the individual as insufficiently active or active.
Eating habits | Baseline (week 0) to post-training (week 13)
  The Food Frequency Questionnaire (FFQ) is used to monitor eating habits. According to the Brazilian Food Guidelines, foods are divided into two groups: in natura/minimally processed foods and processed or ultra-processed foods. The instrument includes a list of 16 foods, and scores are assigned to each based on how often participants report consuming them. The scores can range from 0 to 32 points, with higher scores indicating healthier eating habits. An overall healthy eating score is also calculated by summing all evaluated foods, ranging from 0 to 64 points, where higher scores reflect better eating habits.
Adherence assessments | Intervention period (week 1 to week 12)
  Adherence measures are taken into account for attendance and compliance in interventions. Attendance is monitored through the session's frequency recording and expressed as the percent of intervention sessions experienced by a participant, given the total number of scheduled sessions. Compliance is defined as the percentage of intervention sessions performed without protocol deviations.
Monitoring the intensity of training sessions | Intervention period (week 4, week 8, and week 12).
  The intensity participants perceive at the end of the last class of each mesocycle is recorded using the perceived exertion index. The validated Brazilian Portuguese version of Borg's Category-Ratio 10 scale, adapted by Foster et al. (2001), is used. The scale has values from 0 to 10, anchored to intensities of perceived effort, with 0 being equivalent to no effort (rest) and 10 to maximum effort.
Follow-up questionnaire | Post-training (week 13)
  Each participant answers 14 questions regarding their perception of the intervention using a 7-point Likert scale, in which "1" means "no total agreement" and "7" means "total agreement". The questionnaire is applied post-intervention to assess the participants' perception of safety, enjoyment, motivation, future outlook, benefits for daily life, influence of intervention partners, exercise-related fatigue, satisfaction, self-confidence in physical performance, supervision preference, changes in lifestyle, including physical activity and dietary habits, and main barriers to group participation.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física e Fisioterapia, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be made available by the Trial Coordinator upon reasonable request.

REFERENCES:
- [Background] Foster C, Florhaug JA, Franklin J, Gottschall L, Hrovatin LA, Parker S, Doleshal P, Dodge C. A new approach to monitoring exercise training. J Strength Cond Res. 2001 Feb;15(1):109-15. PMID 11708692
- [Background] Sao-Joao TM, Rodrigues RC, Gallani MC, Miura CT, Domingues Gde B, Godin G. [Cultural adaptation of the Brazilian version of the Godin-Shephard Leisure-Time Physical Activity Questionnaire]. Rev Saude Publica. 2013 Jun;47(3):479-87. doi: 10.1590/s0034-8910.2013047003947. Portuguese. PMID 24346560
- [Background] Brucki SM, Nitrini R, Caramelli P, Bertolucci PH, Okamoto IH. [Suggestions for utilization of the mini-mental state examination in Brazil]. Arq Neuropsiquiatr. 2003 Sep;61(3B):777-81. doi: 10.1590/s0004-282x2003000500014. Epub 2003 Oct 28. Portuguese. PMID 14595482
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Botega NJ, Bio MR, Zomignani MA, Garcia C Jr, Pereira WA. [Mood disorders among inpatients in ambulatory and validation of the anxiety and depression scale HAD]. Rev Saude Publica. 1995 Oct;29(5):355-63. doi: 10.1590/s0034-89101995000500004. Portuguese. PMID 8731275
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] STROOP, J. R. Studies of interference in serial verbal reactions. Journal of Experimental Psychology, v. 18, n. 6, p. 643-662, 1935.
- [Background] de Paula JJ, Costa DS, Miranda DM, Romano-Silva MA. Brazilian version of the Cognitive Failures Questionnaire (CFQ): cross-cultural adaptation and evidence of validity and reliability. Braz J Psychiatry. 2018 Jul-Sep;40(3):312-315. doi: 10.1590/1516-4446-2017-2227. Epub 2017 Dec 11. PMID 29236920
- [Background] Carvalho GA, Caramelli P. Normative data for middle-aged Brazilians in Verbal Fluency (animals and FAS), Trail Making Test (TMT) and Clock Drawing Test (CDT). Dement Neuropsychol. 2020 Jan-Mar;14(1):14-23. doi: 10.1590/1980-57642020dn14-010003. PMID 32206193
- [Background] Ross TP, Calhoun E, Cox T, Wenner C, Kono W, Pleasant M. The reliability and validity of qualitative scores for the Controlled Oral Word Association Test. Arch Clin Neuropsychol. 2007 May;22(4):475-88. doi: 10.1016/j.acn.2007.01.026. Epub 2007 Feb 20. PMID 17317094
- [Background] Schroeder RW, Twumasi-Ankrah P, Baade LE, Marshall PS. Reliable Digit Span: a systematic review and cross-validation study. Assessment. 2012 Mar;19(1):21-30. doi: 10.1177/1073191111428764. Epub 2011 Dec 6. PMID 22156721
- [Background] Alberton CL, Nunes GN, Rau DGDS, Bergamin M, Cavalli AS, Pinto SS. Vertical Ground Reaction Force During a Water-Based Exercise Performed by Elderly Women: Equipment Use Effects. Res Q Exerc Sport. 2019 Dec;90(4):479-486. doi: 10.1080/02701367.2019.1620910. Epub 2019 Jun 11. PMID 31184984